CLINICAL TRIAL: NCT00828984
Title: Polyethylene Glycol for ACF Reduction and Biomarker Modulation in Individuals With CRC Risk
Brief Title: Macrogol 3350-based Oral Osmotic Laxative in Preventing Cancer in Patients at Risk of Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-01113; NCI-2009-01113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 06-8-01; CDR0000632553; N01CN35157 (NIH); NCI06-8-01 (Other: Northwestern University); NWU06-8-01 (Other: DCP); P30CA060553 (NIH)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Adenomatous Polyp; Colorectal Carcinoma
MeSH Terms: conditions — Adenomatous Polyps; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (high-dose PEG 3350) (Experimental): Patients receive high-dose macrogol 3350-based oral osmotic laxative PO QD. Treatment continues for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: macrogol 3350-based oral osmotic laxative; Other: Laboratory Biomarker Analysis
- Arm B (low-dose polyethylene glycol) (Experimental): Patients receive low-dose macrogol 3350-based oral osmotic laxative PO QD. Treatment continues for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: macrogol 3350-based oral osmotic laxative; Other: Laboratory Biomarker Analysis
- Arm C (placebo) (Placebo Comparator): Patients receive placebo PO QD. Treatment continues for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Other: Placebo; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: macrogol 3350-based oral osmotic laxative — Given PO
  Other Names: Colonlytely
  Arms: Arm A (high-dose PEG 3350); Arm B (low-dose polyethylene glycol)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm C (placebo)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well macrogol 3350-based oral osmotic laxative (polyethylene glycol 3350) works in preventing cancer in patients at risk of colorectal cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of macrogol 3350-based oral osmotic laxative may stop cancer from growing in patients who are at risk of colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of polyethylene glycol (PEG) 3350 (administered at 8 g or 17 g/day for six months) versus placebo on epidermal growth factor receptor (EGFR) expression.

SECONDARY OBJECTIVES:

I. To determine the effect of PEG 3350 on aberrant crypt foci (ACF) number and to compare the reduction in ACF number between the low dose (8 g PEG 3350/day) and higher dose (17 g PEG 3350/day) groups.

II. To determine the effect of PEG 3350 on mucosal epithelial proliferation (marker of proliferation Ki-67 [Ki-67]).

III. To determine the effect of PEG 3350 on mucosal apoptosis (cleaved caspase-3).

IV. To determine the effect of PEG 3350 on snail family zinc finger 1 (SNAIL) protein expression.

V. To determine the effect of PEG 3350 on messenger ribonucleic acid (mRNA) expression of SNAIL and EGFR.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients receive high-dose macrogol 3350-based oral osmotic laxative orally (PO) once daily (QD).

ARM B: Patients receive low-dose macrogol 3350-based oral osmotic laxative PO QD.

ARM C: Patients receive placebo (i.e., maltodextrose powder) PO QD.

In all arms, treatment begins within 6-10 days after colonoscopy and continues for up to 6 months in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* History of any size adenoma, known adenoma on present exam, or colon cancer within the last 6 years
* Scheduled for colonoscopy
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to forego PEG laxative during the study period; if the patient has been on a consistent dose of non-PEG laxative for 90 days prior to study entry, the participant may continue those laxatives; participants must agree to restrict additional laxative use to the rescue medication (bisacodyl) provided
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (equivalent to Karnofsky >= 70%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* International normalized ratio (INR) =< 1.5
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X institutional ULN
* Estimated glomerular filtration rate (eGFR) > 45
* Blood urea nitrogen (BUN) < 40
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; restricting intercourse to a surgically sterilized partner; abstinence) for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* If patients are on a dose of cardioprotective aspirin, they must have been on a stable dose for three months prior to colonoscopy and agree to remain at that dose for the six months duration of the study; in addition, patients must agree to limit therapeutic nonsteroidal anti-inflammatory drug (NSAID) use (e.g. pain relief) to no more than 30 cumulative days during the six month duration of the trial

Exclusion Criteria:

* Average of > 2 bowel movements per day for the 90 days preceding study entry as assessed by self-report at baseline
* Average consistency of stools described as watery or loose for the 90 days preceding study entry as assessed by self-report at baseline
* Systemic chemotherapy for any cancer within 18 months prior to enrollment or evidence of active malignant disease
* Radiation to the rectum within 24 months prior to enrollment
* Polyethylene glycol use within 3 months of enrollment (except as part of colonoscopy preparation)
* Systemic corticosteroid use
* Anticoagulant therapy
* Inflammatory bowel disease
* Removal of the rectum
* Evidence of proctitis (radiation, inflammatory bowel disease [IBD], infectious, etc.) by history or endoscopy
* Other investigational agent use within 30 days prior to enrollment
* History of adverse reactions attributed to compounds of similar chemical or biologic composition to polyethylene glycol, bisacodyl or methylene blue
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Patient must not have used suppository medication or enemas for the three months prior to the trial or for the duration of the trial except as directed for colonoscopy or flexible sigmoidoscopy procedure bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Boston Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Wali RK, Bianchi L, Kupfer S, De La Cruz M, Jovanovic B, Weber C, Goldberg MJ, Rodriguez LM, Bergan R, Rubin D, Tull MB, Richmond E, Parker B, Khan S, Roy HK. Prevention of colonic neoplasia with polyethylene glycol: A short term randomized placebo-controlled double-blinded trial. PLoS One. 2018 Apr 4;13(4):e0193544. doi: 10.1371/journal.pone.0193544. eCollection 2018. PMID 29617381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Age 18 and older; Recruitment sites: NorthShore University HealthSystem, University of Chicago, Boston University (no accrual occurred)
Pre-assignment Details: History of any size adenoma or colon cancer within the last 6 years;
Groups:
- Arm A (High-dose PEG 3350): Patients receive high-dose macrogol 3350-based oral osmotic laxative PO QD. Treatment continues for up to 6 months in the absence of unacceptable toxicity.
  17g day/macrogol 3350-based oral osmotic laxative: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Arm B (Low-dose Polyethylene Glycol): Patients receive low-dose macrogol 3350-based oral osmotic laxative PO QD. Treatment continues for up to 6 months in the absence of unacceptable toxicity.
  8g day/macrogol 3350-based oral osmotic laxative: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Started | 28 | 31 | 28
Randomization | 28 | 31 | 28
Treatment | 24 | 26 | 24
Flexible Sigmoidoscopy | 20 | 19 | 19
Post Intervention Follow-Up | 15 | 16 | 19
Completed | 14 | 15 | 19
Not Completed | 14 | 16 | 9
Not completed — Adverse Event | 2 | 3 | 0
Not completed — Lost to Follow-up | 5 | 3 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 4
Not completed — Ineligable | 1 | 2 | 0
Not completed — Medical Contraindication | 0 | 1 | 0
Not completed — Noncompliant | 1 | 2 | 3
Not completed — ConMed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo) | Total
Number analyzed (Participants) | 28 | 31 | 28 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 18 | 55
  >=65 years | 9 | 13 | 10 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 12 | 43
  Male | 14 | 14 | 16 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 27 | 29 | 28 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 0 | 9
  White | 24 | 26 | 26 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference (After Treatment Minus Before Treatment) of EGFR Expression
Description: Evaluate the effect of polyethylene glycol (PEG) 3350 (administered at 8g or 17g/day for six months) versus placebo on EGFR expression.
Time Frame: 6 months - baseline
Population: The study population includes men and women of all races and ethnicities who are scheduled to undergo colonoscopy for a history of colonic neoplasia (within the past 6 years of either colonic adenoma ≥ 5 mm or carcinoma).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
ng/ml | 0.17 (1.07) | -0.40 (0.66) | 0.21 (0.67)

2. Secondary Outcome: Change in ACF Count as Measured in Endoscopically Normal (Non-ACF) Mucosal Biopsies
Description: To determine the effect of PEG 3350 on aberrant crypt foci (ACF) number and to compare the reduction in ACF number between the low dose (8g PEG 3350 / day) and higher dose (17g PEG 3350 / day) groups
Time Frame: 6 months - baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Aberrant Crypt Foci
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
Aberrant Crypt Foci | 2.11 (4.63) | 1 (1.73) | -0.73 (2.74)

3. Secondary Outcome: Change in Ki-67 (Proliferation) Expression as Measured in Endoscopically Normal (Non-ACF) Mucosal Biopsies
Description: To determine the effect of PEG 3350 on mucosal epithelial proliferation (Ki-67)
Time Frame: 6 months - baseline
Population: To determine the effect of PEG 3350 on aberrant crypt foci (ACF) number and to compare the reduction in ACF number between the low dose (8g PEG 3350 / day) and higher dose (17g PEG 3350 / day) groups.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
ng/ml | 2.74 (5.20) | -0.86 (6.62) | -3.58 (11.84)

4. Secondary Outcome: Change in Mucosal Apoptosis (Cleaved Caspase-3) as Measured in Endoscopically Normal (Non-ACF) Mucosal Biopsies
Description: Change in activated caspase-3 (apoptosis) expression as measured in endoscopically normal (non-ACF) mucosal biopsies
Time Frame: 6 months - baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
ng/ml | -0.27 (2.97) | 0.25 (3.18) | -0.15 (2.3)

5. Secondary Outcome: Change in SNAIL Expression as Measured in Endoscopically Normal (Non-ACF) Mucosal Biopsies
Time Frame: 6 months - baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
ng/ml | 0.45 (0.58) | 0.55 (0.88) | 0.08 (0.70)

6. Secondary Outcome: Change in E-cadherin Expression as Measured in Endoscopically Normal (Non-ACF) Mucosal Biopsies
Time Frame: 6 months - baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Number analyzed (Participants) | 14 | 15 | 19
ng/ml | -0.17 (1.75) | 0.15 (0.59) | -0.18 (0.82)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm A (High-dose PEG 3350) | Arm B (Low-dose Polyethylene Glycol) | Arm C (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/31 | 2/28
Other Adverse Events (participants affected / at risk) | 13/28 | 16/31 | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (High-dose PEG 3350) (N=28) | Arm B (Low-dose Polyethylene Glycol) (N=31) | Arm C (Placebo) (N=28)
Hemorrgae/Bleeding,CNS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Perforation,GI: Colon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (High-dose PEG 3350) (N=28) | Arm B (Low-dose Polyethylene Glycol) (N=31) | Arm C (Placebo) (N=28)
Edema; Limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, GI: Rectum (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrythmia: Supraventricular and nodal arrhythmia: Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otitis, Middle Ear (Non-Infectious) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis, External Ear (Non-Infectious) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine - Other (Specify, __) (Endocrine disorders) | 8 (17) | 1 (1) | 0 (0) — Pancreatic Cancer
Diarrhea (Gastrointestinal disorders) | 8 (8) | 4 (5) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (8) | 2 (2) | 3 (4)
Distention/bloating, Abdominal (Gastrointestinal disorders) | 6 (13) | 3 (4) | 3 (5)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal - Other (Specify) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) — Urgency to have bowel movement
Pain: Pain Nos (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 0 (0) | 1 (4) | 0 (0) — Sinus Headache Side Pain Body Ache Abdominal Pain
Pain: Muscle (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain: Abdomen Nos (General disorders) | 2 (6) | 1 (1) | 4 (6)
Pain: Joint (General disorders) | 0 (0) | 1 (2) | 2 (8)
Pain: Neuralgia/Peripheral Nerve (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain: Throat/Pharynx/Larynx (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain: Stomach (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain: Rectum (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain: Chest/Thorax Nos (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain: Back (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain: Dental/Teeth/Peridontal (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain: Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
"Constitutional Symptoms: Fever (In the absence of Neutropenia, where Neutropenia is defined as ANC (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constitutional Symptoms: Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syndromes: Flu-like Syndrome (General disorders) | 0 (0) | 2 (6) | 0 (0)
Allergic Rhinitis (Including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 2 (2) | 2 (2)
Infection with normal ANC or Grade 1 or 2 Neutrophils: Nerve-Peripheral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC: Upper Airway Nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Recurrent Skin Boil
Infection with unknown ANC: Pharynx (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 Neutrophils: Upper Airway Nos (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Infection with unknown ANC: Skin (Cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
"Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils (ANC <1.0 X 1 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Nerve-Peripheral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Dental-tooth (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Sinus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC: Bladder (Urinary) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal/Soft tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Plantar Fascitis
Musculoskeletal/Soft tissue - Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary/Upper Respiratory: Nasal Cavity/Paranasal Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory: Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less